CLINICAL TRIAL: NCT02472639
Title: Impact of Ostom-i Alert Sensor on Quality of Life in Patients With Ileostomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient compliance issues
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Karen Zaghiyan, Colon & Rectal Surgeon, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00040251
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Results first posted 2017-10-03 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Ostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ostom-i Alert Sensor (Experimental): Patients will wear Ostom-i sensor
  Interventions: Device: Ostom-i Alert Sensor
- No Ostom-i Alert Sensor (Other): Patient will not wear Ostom-i sensor
  Interventions: Other: No Ostom-i Alert Sensor

INTERVENTIONS:
Device: Ostom-i Alert Sensor — Wear the Ostom-i Alert Sensor
  Arms: Ostom-i Alert Sensor
Other: No Ostom-i Alert Sensor — Patient will not use device
  Arms: No Ostom-i Alert Sensor

SUMMARY:
The purpose of this study is to evaluate patient satisfaction and quality of life in patients with ileostomy managed with or without the novel Ostom-i Alert device.

DETAILED DESCRIPTION:
Patients with ileostomy have impaired quality of life related to their ileostomy (Person et al. DCR. 2012; 55: 783 - 787; Scarpa et al. Colorectal Dis. 2010; 12: 914 - 920). Although patients with ileostomy have better overall quality of life compared with colostomy patients (Silva et al. Worl J Surg. 2003; 27: 421-424), the liquid nature of the ileostomy effluent predisposes these patients to bag overfilling and dehydration more so than colostomy patients (Paquette et al. DCR 2013; 56: 974-979). This may be specifically important in populations with long term or permanent ileostomy. Overfilling and breakage/leakage of the ileostomy bag can also affect patient's ability to function in social environments, go out in public, have intimate relationships with significant others, and interfere with sleep patterns (due to high output and nighttime overfilling of the ileostomy bag).

The Ostom-i Alert is a novel device developed by a patient with ileostomy and now FDA approved in the United States. The device is a sensor that clips onto any ostomy bag and sends a Bluetooth signal to a mobile device app. An alarm lets the patient know before the stoma bag is at risk for overfilling and leaking. The potential advantage is that the device can prevent unexpected bag overfilling, breakage, and nighttime accidents. This may therefore lead to improved quality of life. The volume and output recordings can also be stored and emailed to the patient's health care providers, with potential to reduce ostomy related dehydration through more accurate volume recording and sharing.

While the device has many applications, the purpose of this research study is to specifically evaluate patient quality of life after application of the Ostom-i Alert compared with standard ostomy care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ileostomies in place without a plan for ileostomy take down in the next 4 months.
2. Able to freely give written informed consent to participate in the study and have signed the Informed Consent Form;
3. Males or females, age 18 and older at the time of study screening;
4. Patients with loop or end ileostomy at least 1 month since ileostomy creation
5. No plan for stoma reversal for the next 4 months to allow adequate time for study inclusion
6. Patients who own an iPhone, iPod Touch, or Android device

Exclusion Criteria:

1. Mentally incompetent or unable or unwilling to provide informed consent or comply with study procedures;
2. Children <18
3. Pregnant patients
4. Patients with planned ileostomy closure in the next 4 months
5. Patients with colostomy, more than one ostomy, or urostomy
6. Patients unable or unwilling to come in for in person Ostomi-I Alert teaching and screening visits
7. Patients without an iPhone, iPod Touch, or Android device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-06-10 (Actual); Primary Completion 2016-05-26 (Actual); Study Completion 2016-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Zaghiyan, MD, Principal Investigator — Cedars-Sinai Medical Center

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
Started | 4 | 3
Completed | 0 | 0
Not Completed | 4 | 3
Not completed — Physician Decision | 4 | 3

BASELINE CHARACTERISTICS:
Population: Study was prematurely terminated. Data was not collected or analyzed due to issue with study compliance.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Patient Quality of Life as Measured by the 20-item Stoma-QOL Questionnaire at 1 Month and 3 Month Follow-up After Using the Ostomi-I Alert Versus Standard Stoma Care Without the Ostom-i Alert.
Time Frame: up to 3 Months
Population: Study was prematurely terminated. Data was not collected or analyzed due to issue with study compliance.
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Satisfaction With Ostom-i Device
Description: Study was prematurely terminated. Data was not collected or analyzed due to issue with study compliance.
Time Frame: 3 months
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Ostomy Bag Breakages During the Study Period
Description: Study was prematurely terminated. Data was not collected or analyzed due to issue with study compliance.
Time Frame: 3 months
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Score on Additional QOL Questions Not Included in Stoma-QoL Questionnaire
Description: Study was prematurely terminated. Data was not collected or analyzed due to issue with study compliance.
Time Frame: 3 months
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Dehydration Related Hospital Admissions During Study Period
Description: Study was prematurely terminated. Data was not collected or analyzed due to issue with study compliance.
Time Frame: 3 months
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data were not collected and no data was analyzed. Study was terminated due to issues with compliance and enrollment. Total number of participants at Risk (e.g., "All-Cause Mortality, Serious, and other[ Not Including Serious] adverse events were not monitored/assessed for this study.
Arm/Group | Ostom-i Alert Sensor | No Ostom-i Alert Sensor
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Study only accrued 7 patients. Due to non-compliance and issues with the device it was decided to terminate the study.

No data analysis has been done and will not be done in the future. This study was been closed with the IRB.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No